CLINICAL TRIAL: NCT02485769
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo Controlled, Sequential Group, Multiple Ascending Dose Escalation Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Orally Administered Pf 06650833 In Healthy Subjects
Brief Title: Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Oral Pf-06650833 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: B7921002; IRAK4 MAD (Other: Alias Study Number)
Record Dates: First submitted 2015-05-28; First posted 2015-06-30 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06650833 (Experimental): Active arm , PF-06650833 kinase.
  Interventions: Drug: PF-06650833
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06650833 — Suspension
  Arms: PF-06650833
Drug: Placebo — Suspension
  Arms: Placebo
Drug: PF-06650833 — Tablet (Modified Release)
  Arms: PF-06650833
Drug: Placebo — Tablet (Modified Release)
  Arms: Placebo

SUMMARY:
A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo Controlled, Sequential Group, Multiple Ascending Dose Escalation Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Orally Administered PF-06650833 In Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non childbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
5. Smokers must not exceed the equivalent of 5 cigarettes per day.
6. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
7. Screening supine blood pressure100 mm Hg (systolic) or 50 mm Hg (diastolic); or 140 mm Hg (systolic) or 90 mm Hg (diastolic) following at least 5 minutes of supine rest. If blood pressure (BP) is 40 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
8. Screening pulse or heart rate (HR) >100 bpm after at least 5 minutes of rest. If the pulse/HR is >100 bpm, the pulse/HR should be repeated two more times (separated by at least 2 minutes) and the average of the three pulse/HR values should be used to determine the subject's eligibility.
9. Screening 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
10. Clinically significant abnormality on chest X ray performed at screening or within 3 months of screening date.
11. History of tuberculosis or active or latent or inadequately treated infection, positive Quantiferon TB test
12. History of hepatitis or HIV, positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HepBsAg), hepatitis B core antibodies (HepBcAb) or hepatitis C antibodies (HCVAb).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events. | 50 days
Incidence and Magnitude of Participants with Treatment-emergent hematology clinical abnormalities | 50 days
Incidence and Magnitude of Participants with Treatment-emergent chemistry abnormalities (including, cardiac enzymes CK, CK-MB and cardiac Troponin-1, serum myoglobin) | 50 days
Incidence and Magnitude of Participants with Treatment-emergent urinalysis abnormalities | 50 Days
Changes from baseline in blood pressure | 50 days
Changes from baseline in pulse rate | 50 days
Changes from baseline in respiratory rate | 50 days
Changes from baseline in ECG parameters (standard 12-lead ECG) | 50 days
Changes from baseline in Epstein-Barr virus [EBV] | 50 days
Changes from baseline in Cytomegalovirus [CMV] | 50 days
Changes from baseline in Herpes simplex virus-1 and -2 [HSV-1 and HSV-2] | 50 days

SECONDARY OUTCOMES:
To characterize Cmax in plasma | Day 1 and Day 14
To determine PF-06650833 excreted unchanged (AE tau and AE tau %), | Day 14
To characterize Tmax in plasma | Day 1 and Day 14
To characterize AUC tau in plasma | Day 1 and Day 14
To characterize Cmin in plasma | Day 1 and Day 14
Characterize Cmax (dose normalized) in plasma | Day 1 and Day 14
To characterize AUC tau(dose normalized) in plasma | day1 and day 14
To determine the renal clearance (CLr) | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Winkler A, Sun W, De S, Jiao A, Sharif MN, Symanowicz PT, Athale S, Shin JH, Wang J, Jacobson BA, Ramsey SJ, Dower K, Andreyeva T, Liu H, Hegen M, Homer BL, Brodfuehrer J, Tilley M, Gilbert SA, Danto SI, Beebe JJ, Barnes BJ, Pascual V, Lin LL, Kilty I, Fleming M, Rao VR. The Interleukin-1 Receptor-Associated Kinase 4 Inhibitor PF-06650833 Blocks Inflammation in Preclinical Models of Rheumatic Disease and in Humans Enrolled in a Randomized Clinical Trial. Arthritis Rheumatol. 2021 Dec;73(12):2206-2218. doi: 10.1002/art.41953. Epub 2021 Nov 1. PMID 34423919
- [Derived] Danto SI, Shojaee N, Singh RSP, Li C, Gilbert SA, Manukyan Z, Kilty I. Safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06650833, a selective interleukin-1 receptor-associated kinase 4 (IRAK4) inhibitor, in single and multiple ascending dose randomized phase 1 studies in healthy subjects. Arthritis Res Ther. 2019 Dec 5;21(1):269. doi: 10.1186/s13075-019-2008-6. PMID 31805989
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7921002&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double%20Blind%2C%20Sponsor%20Open%2C%20Placebo%20Controlled%2C%20Sequential%20Group%2C%20Multiple%20Ascending%20Dose%20Escalation%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20Orally%20Administered%20Pf%2006650833%20In%20Healthy%20Subjects